CLINICAL TRIAL: NCT05280496
Title: Implementation of a Pragmatic Approach to Lower Diabetes Mellitus Risk After a Diagnosis of Gestational Diabetes Mellitus
Brief Title: A Pragmatic Approach to Lower Diabetes Risk After Gestational Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002576
Record Dates: First submitted 2022-03-03; First posted 2022-03-15 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-09

CONDITIONS: Diabetes, Gestational; PreDiabetes; Diabetes Mellitus, Type 2
Keywords: gestational diabetes; diabetes risk; medical management; risk prevention; postpartum; diabetes; metformin
MeSH Terms: conditions — Diabetes, Gestational; Prediabetic State; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Metformin (Experimental): Participants will be given a daily prescription of metformin for 12 months postpartum. At 12 months and again at 15 months (3 months off the drug), HbA1c and weight will be assessed.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is used to lower blood sugar in patients with high blood sugar (diabetes).

SUMMARY:
This study is testing whether daily metformin for 1 year postpartum can reduce risk of diabetes in patients who had gestational diabetes. Typical care for prediabetes after gestational diabetes is counseling on diet and lifestyle. This study is researching whether management of diabetes prevention is more effective with the drug metformin. This study will be conducted at Tufts Medical Center.

DETAILED DESCRIPTION:
Women with a history of gestational diabetes mellitus (GDM) represent a unique population who may benefit from metformin as much as lifestyle intervention; when metformin is prescribed to these women remote from delivery after a diagnosis of prediabetes, it reduces their risk of developing diabetes mellitus (DM) by up to 40% over 10 years. However, in the current system in which gestational diabetes diagnosis, prediabetes testing, and metformin prescription are temporally separated by months to years, less than 20% of postpartum women undergo prediabetes testing. When prediabetes is identified in women with a history of GDM, only 7.8% are prescribed metformin.

Given the increasing public health burden of DM, there is an urgent need to remedy this problem and correct this deficiency in health care delivery that allows so many at-risk women to remain unidentified and untreated.

Compelling preliminary data, confirmed at several other sites, indicates that the postpartum glucose tolerance test to identify individuals with prediabetes can be moved from 4-12 weeks postpartum to 1-4 days postpartum, when women are still hospitalized, with test compliance of 92% and no reduction in sensitivity or specificity for prediabetes.

When individuals with a history of GDM and prediabetes are prescribed metformin, they experience a 50% reduction in DM risk and a 3 kg increase in weight loss over three years compared to placebo. If these same benefits are realized when metformin is initiated soon after delivery, then a simple change in postpartum care so that metformin is routinely prescribed at hospital discharge to women with a history of GDM and prediabetes could improve the health of thousands of women annually by decreasing the number of women who develop DM and fail to achieve postpartum weight loss.

Each year in the United States, approximately 280,000 women are diagnosed with GDM. Without intervention, up to 70% of these women will develop diabetes mellitus (DM) over their lifetime, resulting in devastating health consequences and escalating health care costs. However, implementing a postpartum glucose tolerance test and intervening with metformin for those with prediabetes may be a cost-effective change to postpartum care that would result in a profound decrease in DM incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Women currently pregnant with planned delivery at Tufts Medical Center
2. Gestational diabetes mellitus diagnosed during pregnancy
3. ≥18 years of age
4. Opted for the 2 hour 75 gram OGTT during postpartum hospitalization
5. Willing and able to sign the informed consent

Exclusion Criteria:

1. Unable to commit to required study visits for any reason.
2. Contraindications to metformin

   * Liver disease
   * Impaired renal function (Creatinine Clearance> )
   * Congestive heart failure(CHF)
   * Taking drugs that could interfere with metformin metabolism
3. Taking metformin outside of pregnancy
4. Prescribed medications for chronic disease that affect glucose metabolism (e.g., long term oral steroids).
5. Decided against the 2 hour 75 gram OGTT during postpartum hospitalization.
6. Preexisting diabetes mellitus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
HbA1C | 12 months
  These results will be shared with participants and their providers. Any participants who accepted metformin but do not have diabetes will be asked to stop all study medication and no more study medication will be dispensed.
HbA1C | 15 months
  At 15 months postpartum, study participants with prediabetes will be seen again for their final study visit. The investigators intend to follow all participants for 3 months after metformin treatment ends for both safety reasons and efficacy reasons. If the metformin was masking diabetes, the investigators want the opportunity to identify those participants and refer them for treatment. Additionally, prior studies have not determined whether the benefits of metformin extend after the medication is discontinued (as indicated by the FDA when the investigators requested to use metformin in the first year postpartum).

SECONDARY OUTCOMES:
Weight | 12 months
Weight | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Erika Werner, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charlton JM, van Heyningen R. Glucose 6-phosphate dehydrogenase in the mammalian lens. Exp Eye Res. 1971 Mar;11(2):147-60. doi: 10.1016/s0014-4835(71)80018-0. No abstract available. PMID 4399293
- [Background] Carter EB, Tuuli MG, Odibo AO, Macones GA, Cahill AG. Prenatal visit utilization and outcomes in pregnant women with type II and gestational diabetes. J Perinatol. 2017 Feb;37(2):122-126. doi: 10.1038/jp.2016.175. Epub 2016 Oct 13. PMID 27735930
- [Background] Dinglas C, Muscat J, Heo H, Islam S, Vintzileos A. Immediate Postpartum Glucose Tolerance Testing in Women with Gestational Diabetes: A Pilot Study. Am J Perinatol. 2017 Oct;34(12):1264-1270. doi: 10.1055/s-0037-1606620. Epub 2017 Sep 14. No abstract available. PMID 28910846
- [Background] Asymptomatic hiatus hernia. Lancet. 1969 Apr 26;1(7600):870-1. No abstract available. PMID 4180530
- [Background] Moin T, Li J, Duru OK, Ettner S, Turk N, Keckhafer A, Ho S, Mangione CM. Metformin prescription for insured adults with prediabetes from 2010 to 2012: a retrospective cohort study. Ann Intern Med. 2015 Apr 21;162(8):542-8. doi: 10.7326/M14-1773. PMID 25894024
- [Background] Ratner RE, Christophi CA, Metzger BE, Dabelea D, Bennett PH, Pi-Sunyer X, Fowler S, Kahn SE; Diabetes Prevention Program Research Group. Prevention of diabetes in women with a history of gestational diabetes: effects of metformin and lifestyle interventions. J Clin Endocrinol Metab. 2008 Dec;93(12):4774-9. doi: 10.1210/jc.2008-0772. Epub 2008 Sep 30. PMID 18826999
- [Background] Werner EF, Has P, Rouse D, Clark MA. Two-day postpartum compared with 4- to 12-week postpartum glucose tolerance testing for women with gestational diabetes. Am J Obstet Gynecol. 2020 Sep;223(3):439.e1-439.e7. doi: 10.1016/j.ajog.2020.05.036. Epub 2020 May 26. PMID 32470456
- [Background] Werner EF, Has P, Kanno L, Sullivan A, Clark MA. Barriers to Postpartum Glucose Testing in Women with Gestational Diabetes Mellitus. Am J Perinatol. 2019 Jan;36(2):212-218. doi: 10.1055/s-0038-1667290. Epub 2018 Jul 30. PMID 30060291
- [Background] Werner EF, Has P, Tarabulsi G, Lee J, Satin A. Early Postpartum Glucose Testing in Women with Gestational Diabetes Mellitus. Am J Perinatol. 2016 Aug;33(10):966-71. doi: 10.1055/s-0036-1583193. Epub 2016 Apr 27. PMID 27120481
- [Background] Whelan AR, Ayala NK, Werner EF. Postpartum Use of Weight Loss and Metformin for the Prevention of Type 2 Diabetes Mellitus: a Review of the Evidence. Curr Diab Rep. 2021 Sep 8;21(10):37. doi: 10.1007/s11892-021-01410-7. PMID 34495405
- [Background] Bennett WL, Liu SH, Yeh HC, Nicholson WK, Gunderson EP, Lewis CE, Clark JM. Changes in weight and health behaviors after pregnancies complicated by gestational diabetes mellitus: the CARDIA study. Obesity (Silver Spring). 2013 Jun;21(6):1269-75. doi: 10.1002/oby.20133. Epub 2013 May 13. PMID 23666593
- See also: The Diabetes Prevention Program — https://doi.org/10.2337/diacare.25.12.2165